CLINICAL TRIAL: NCT05773989
Title: Pharmacodynamic Outcomes in Patients With Coronary Artery Disease Undergoing Percutaneous Coronary Intervention Treated With an Individualized Treatment STRATEGY
Brief Title: Pharmacodynamic Outcomes in CCS Patients Treated With an Individualized Treatment Strategy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, Principal Investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-504078-39
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Platelet Reactivity
Keywords: Percutaneous Coronary Intervention; Antithrombotic therapy; CYP2C19; CYP2C19 guided treatment; Pharmacodynamics
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Prasugrel Hydrochloride; Clopidogrel; Aspirin

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotype guided P2Y12 monotherapy (Experimental): Patients will be tested for the CYP2C19 genotype. Patients without a loss-of-function (LOF) allele will receive clopidogrel monotherapy (tablet of 75mg once daily) for 6 months. Patients with a LOF-allel will receive ticagrelor (tablet of 90mg twice daily) or prasugrel (tablet of 10mg once daily) for 6 months.
  Interventions: Drug: CYP2C19 genotype guided P2Y12 monotherapy
- Standard DAPT (Active Comparator): Patients will receive clopidogrel monotherapy (tablet of 75mg once daily) for 6 months and acetylsalicylic acid (tablet 80mg one daily) for 6 months.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: CYP2C19 genotype guided P2Y12 monotherapy — Patients without a LOF-allel will receive clopidogrel monotherapy (tablet of 75mg once daily) for 6 months. Patients with a LOF-allel will receive ticagrelor (tablet of 90mg twice daily) or prasugrel (tablet of 10mg once daily) for 6 months.
  Other Names: Ticagrelor; Prasugrel; Clopidogrel
  Arms: Genotype guided P2Y12 monotherapy
Drug: Clopidogrel — Standard DAPT according to current guidelines with clopidogrel (tablet of 75mg once daily) for 6 months and acetylsalicylic acid (tablet 80mg one daily) for 6 months.
  Other Names: Aspirin
  Arms: Standard DAPT

SUMMARY:
Patients with Chronic Coronary Syndrome (CCS) undergoing with elective percutaneous coronary intervention (PCI) are treated with dual antiplatelet therapy (DAPT), consisting of aspirin combined with clopidogrel for 6 months. The aim of DAPT is to prevent recurrent thrombotic events, i.e. death, stent thrombosis and/ or myocardial infarction (MI). However, the trade-off of thrombotic prevention by DAPT is an increased risk of bleeding.

Multiple strategies to reduce bleeding risk and optimize outcomes have been proposed. On one hand the bleeding risk can be reduced by shortening the duration of DAPT and omitting aspirin. This has been proven effective in patients with acute coronary syndromes (ACS) compared to standard DAPT, without a significant difference in thrombotic events. On the other hand, personalized medicine by means of genotyping to ensure that a patient is treated with an, for them, effective drug, can be a strategy to optimize patients outcomes. In CCS patients the preferred P2Y12-inhibitor is clopidogrel. However, clopidogrel must first be activated by the CYP2C19 enzyme in the liver. Only then can clopidogrel inhibit the P2Y12-receptor and prevent platelet activation. Almost thirty percent of patients has a genetic variation of the gene encoding this CYP2C19 enzyme. In these patients, clopidogrel is not or hardly activated, putting them at a higher risk of thrombotic events than patients who do not have this gene variation. By determining the CYP2C19 genotype, it is possible to estimate whether clopidogrel will be effective or not.

In this trial the investigators evaluate the pharmacodynamic effects of genotype guided P2Y12-inhibitor monotherapy in patients with CCS undergoing PCI. In the intervention arm the CYP2C19 genotype will be assessed using a point-of-care test device on the cardiology ward, which can be performed by (research) nurses. Patients with a CYP2C19 loss-of-function (LOF) allel will be treated with monotherapy ticagrelor or prasugrel. Patients who are non-carrier of a LOF allel will receive clopidogrel. The control arm will be treated with the current standard-of-care, which is DAPT, consisting of aspirin combined with clopidogrel for 6 months.

The main goals is to assess the antithrombotic effects of individualized P2Y12 monotherapy strategy versus clopidogrel plus aspirin in elective PCI patients.

DETAILED DESCRIPTION:
Rationale: Novel antithrombotic strategies, such as genotype-guided P2Y12-inhibitor selection and P2Y12-inhibitor monotherapy, instead of routine dual antithrombotic therapy (DAPT), have recently been investigated in major randomized controlled trials. It is unclear whether these therapies can also be applied to all comer patients undergoing elective percutaneous coronary (PCI) with stenting.

Objective: The aim of this study is to evaluate the pharmacodynamic response of CYP2C19-genotype-guided monotherapy in patients undergoing elective PCI. Bleeding and ischemic outcomes will also be registered.

Study design: A prospective, single center, randomized controlled trial.

Study population: Patients undergoing elective PCI

Intervention: Randomized to genotype-guided monotherapy P2Y12 inhibition or standard DAPT.

After PCI, patients will be randomised between two groups. Intervention group: P2Y12-inhibitor monotherapy. Patients without a LOF-allel will receive clopidogrel monotherapy (tablet of 75mg once daily) for 6 months. Patients with a LOF-allel will receive ticagrelor (tablet of 90mg twice daily) or prasugrel (tablet of 10mg once daily) for 6 months.

Control group: Dual antiplatelet therapy (DAPT). Patients will receive clopidogrel (tablet of 75mg once daily) for 6 months and acetylsalicylic acid (tablet 80mg one daily) for 6 months.

Main study parameters/endpoints:

• To evaluate the antithrombotic effects of ticagrelor/prasugrel or clopidogrel monotherapy versus clopidogrel plus aspirin in order to assess the feasibility and safety of individualized antithrombotic therapy after elective PCI based on CYP2C19-genotyping.

Secondary endpoints:

* The primary (safety) bleeding endpoint is the incidence of minor, moderate or severe bleeding (Bleeding Academic Research Consortium 2, 3 and 5)
* The primary efficacy endpoint is the incidence of cardiovascular mortality, myocardial infarction, stent thrombosis, and stroke)
* Individual components and combinations of the primary and secondary end points
* To evaluate the net clinical benefit (a composite of all-cause death, MI, stroke and major bleeding defined as BARC type 3 or 5 bleeding at 6 months)
* To compare the number of patients in whom the antiplatelet drug is prematurely discontinued or switched to another drug in the CYP2C19 genotype guided antiplatelet treatment versus standard DAPT treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Patients with CCS undergoing successful elective PCI
* Patients with written informed consent as approved by the ethics committee

Exclusion Criteria:

* Contraindication to aspirin, ticagrelor, prasugrel or clopidogrel
* Under the age of 18 years
* Planned cardiac valve surgery
* Need for chronic oral anticoagulation
* PCI when admitted for ACS
* Life expectancy < 1 year
* Unable or unwilling to provide informed consent
* Pregnancy
* Suboptimal result of stenting as defined by the operator, preferably explained according the complex-PCI criteria
* Treatment with a strong CYP3A4 inhibitor or inducer
* Treatment with a strong CYP2C19 inhibitor or inducer
* History of definite stent thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity | Baseline and 30 days after PCI
  Change in P2Y12 Reaction Units (PRU) measured using the VerifyNow
High on-treatment platelet reactivity (HTPR) | 30 days
  Number of participants with high on-treatment platelet reactivity (HTPR) defined by a PRU >208

SECONDARY OUTCOMES:
Bleeding complications | 6 months
  Number of participants with major or clinically relevant bleeding complications according to the Bleeding Academic Research Consortium Definition for Bleeding (BARC) classification.
Myocardial infarction | 6 months
  Number of participants with myocardial infarction as defined by the 4th Universal Definition of Myocardial Infarction
Stroke | 6 months
  Number of participants with stroke as defined by the Valve Academic Research Consortium (VARC) definitions
Stent thrombosis | 6 months
  Number of participants with stent thrombosis as defined by the Academic Research Consortium (ARC)
All-cause death | 6 months
  Number of participants with all-cause death as defined by the Academic Research Consortium (ARC)
Cardiovascular death | 6 months
  Number of participants with cardiovascular death as defined by the Academic Research Consortium (ARC)

CONTACTS AND LOCATIONS:
Overall Officials: Jurriën ten Berg, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No